CLINICAL TRIAL: NCT05590416
Title: An Observational Study of Adalimumab in the Treatment of Acute Vogt-Koyanagi-Harada Disease
Brief Title: A Study of Adalimumab in Acute Vogt-Koyanagi-Harada Disease
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Xiaomin Zhang, Principal Investigator, MD, PhD, Tianjin Medical University
Other Study IDs: 2022KY-16
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Vogt-Koyanagi-Harada Disease; Adalimumab
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- adalimumab group: The initial dose of glucocorticoid is 1 mg/kg/day, and gradually stops within 90-180 days. Adalimumab is administered subcutaneously at an initial loading dose of 80 mg, followed by a 40 mg dose every other week (q2w) starting from the second week. Therapy will be continued 6 months after the disappearance of active ocular inflammation. Then, injection will extend for 3 days until withdrawal after 40 days apart.
  Interventions: Drug: Adalimumab
- traditional therapy group: Acute VKH patients treatment with only glucocorticosteroid or glucocorticosteroid combined with immunosuppressive agents.

INTERVENTIONS:
Drug: Adalimumab — Adalimumab is administered subcutaneously at an initial loading dose of 80 mg, followed by a 40 mg dose every other week (q2w) starting from the second week. Therapy will be continued 6 months after the disappearance of active ocular inflammation. Then, injection will extend for 3 days until withdrawal after 40 days apart.
  Groups: adalimumab group

SUMMARY:
This project is designed to test the hypothesis that adalimumab is clinically useful for patients with acuta Vogt-Koyanagi-Harada disease

DETAILED DESCRIPTION:
Approval of the study was obtained from the hospital's ethical committee. The study design and methodology followed the tenets of Declaration of Helsinki. All patients were provided with written informed consent and received a thorough explanation of the use of adalimumab, its potential risks and benefits. This is a monocenter, cohort, observational study evaluating patients with acute VKH divided into two groups: adalimumab therapy group and traditional therapy group.

For adalimumab therapy group, an initial dose of 80 mg adalimumab was administered subcutaneously followed by a maintenance dose of 40 mg every two weeks, and data will be collected prospectively with regard to ophthalmologic outcomes. For the traditional therapy group, patients were treated with glucocorticoids alone or glucocorticoids combined with immunosuppressants. Study participants will be followed for up to one year to determine efficacy and side effects.

According to best corrected visual acuity (BCVA), anterior chamber and vitreous inflammation, optical coherence tomography (OCT), change in corticosteroid dose during the study period and so on. The investigators evaluate the anti-inflammatory and immunosuppressive effects of adalimumab in treatment of acute VKH.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 to 70 years of age.
2. Subjects who do not have previous, active or latent tuberculosis (TB).
3. Subject must have Vogt-Koyanagi-Harada disease less than one month.
4. Subject who were previously treated with systemic glucocorticoid less than one week.
5. Subject meets at least 1 of the following criteria:

1)patients who reject using systemic glucocorticoid because of the long-term side effects. 2)patients with other high-risk or systemic disease were limited by the use of glucocorticoid. 3)patients with a little reparation of retinal detachments after a week treatment with powerful systemic glucocorticoid(≥1mg/kg/day).

Exclusion Criteria:

1. Subject with confirmed or suspected infectious uveitis, including but not limited to infectious uveitis due to TB, cytomegalovirus (CMV), Human T-Lymphotropic Virus Type 1 (HTLV-1), Whipple's disease, Herpes Zoster virus (HZV), Lyme disease, toxoplasmosis and herpes simplex virus (HSV).
2. Subject with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial.
3. Subject has previous exposure to anti-tumor necrosis factor (TNF) therapy or any biologic therapy with a potential therapeutic impact on non-infectious uveitis.
4. Subject has received Ozurdex® (dexamethasone implant) within 6 months prior to the Baseline visit.
5. Subject has received intravitreal anti-VEGF therapy within 45 days of the Baseline visit for Lucentis® (ranibizumab) or Avastin® (bevacizumab) or within 60 days of the Baseline visit for anti-VEGF Trap (aflibercept).
6. Subject has received intravitreal methotrexate within 90 days prior to the Baseline visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VKH patients were recruited from the uveitis centre of Tianjin Medical University Eye Hospital
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change In LogMAR Best Corrected Visual Acuity (BCVA) From Baseline to Each Visit. | 24 weeks
  The participant's best corrected visual acuity was measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart. On the logMAR scale, 0 is equivalent to 20/20 visual acuity, the range of normal vision is considered to be from -0.2 - 0.1; higher values indicate visual impairment.
Recurrence rate | 24 weeks
  The recurrence rates in adalimumab treatment group and control group

SECONDARY OUTCOMES:
Change in Anterior Chamber (AC) Cell Grade From Baseline to Each Visit | 24 weeks
  Slit lamp examinations were conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm × 1 mm slit beam was used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria:
  Grade 0 = < 1 cell Grade 0.5+ = 1 - 5 cells Grade 1+ = 6 - 15 cells Grade 2+ = 16 - 25 cells Grade 3+ = 26 - 50 cells Grade 4+ = > 50 cells.
Prednisone exposure | 12 months
  Cumulative prednisone dose and/or mean prednisone dose

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China